CLINICAL TRIAL: NCT04752605
Title: Effectiveness of Play-Based Training on Executive Functioning in Pre-School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Niilo Mäki Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4-C7291
Record Dates: First submitted 2021-01-26; First posted 2021-02-12 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Executive Function; Problem Behavior
Keywords: Preschool; Self-regulation; Executive function; Problem behavior; Training; Play-based
MeSH Terms: conditions — Problem Behavior; Self-Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): play sessions included as a part of normal early childhood education; parents' evening for all parents; parents' group for the parents of children that have difficulties in self-regulation and that are offered more individualized small group activity
  Interventions: Behavioral: Finnish ENGAGE together
- Control (No Intervention): normal early childhood education

INTERVENTIONS:
Behavioral: Finnish ENGAGE together — Early childhood education workers play games with children during day care. The games (e.g. ball games, puzzles, Simon says) target children's executive functions and self-regulatory skills, e.g. inhibition, attention, and emotion regulation. The first phase of the intervention (6 weeks) includes play sessions (15 minutes each day) for all children as well as a parents' evening to encourage playing at home. In the second phase (8 weeks), more individualized small group play sessions (3 times a week, 30 minutes at once) are arranged for the children that show difficulties in self-regulation after the first phase. Also, a parents' group including 6 group sessions and 2 phone calls is arranged for their parents in this phase. The participating parents are asked to play the games for 20 minutes each day with their children. During the group meetings, the parents share their experiences of playing at home and receive support and guidance from 2 health care professionals.
  Arms: Intervention

SUMMARY:
The aim of this study is to examine the effectiveness of a play-based intervention designed to support the development of executive functioning in 3-5-year-old children. The intervention is implemented in the day care setting as a part of early childhood education in collaboration with parents and local healthcare and social welfare workers. The study hypothesizes that the intervention as an add-on to normal early childhood education brings added benefits to the development of children's executive functioning in comparison to early childhood education without the add-on.

DETAILED DESCRIPTION:
This cluster-randomized controlled trial examines the effectiveness of a play-based intervention, added as a component to normal early childhood education, in supporting the development of executive functioning in 3-5-year-old children in comparison to early childhood education without such a component. 12 day care centers in Finland have been randomized to intervention (n = 6) and control (n = 6) groups. The children in the intervention group will receive the intervention in the spring of 2021, and the children in the control group will be on the wait list and receive the intervention in the fall of 2021 after measurements. In the day care centers belonging to the intervention group, play sessions supporting the development of children's executive functioning will be arranged as a part of normal early childhood education. The pre-selected games target children's executive functions and self-regulatory abilities, e.g. inhibition, attention, working memory and emotion regulation. The first phase of the intervention (6 weeks) includes play sessions for all children as well as a parents' evening. In the second phase (8 weeks), more individualized play sessions are arranged for the children that exhibit difficulties in executive functions after the first phase. Also, a parents' group is arranged in this phase, which will expand the daily play activities to homes. Day care education personnel and parents fill out questionnaires concerning children's behavior at 4 time points, and the children participating in the second phase (small group activity) will complete two iPad tasks before and after the small group activity. The study takes place in Finland.

ELIGIBILITY:
Inclusion Criteria:

* Children born between 4.6.2015 - 11.1.2018
* For the second phase (small group activity): children must exhibit problems in executive functions (e.g. inattention, hyperactivity, impulsivity) and be considered as potentially benefitting from additional practice as assessed by early childhood educators

Exclusion Criteria:

-

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
School Situations Questionnaire | Change from baseline at 1,5, 4, and 7 months
  Early childhood education workers assess whether children exhibit problem behaviors in different preschool situations and the severity of the problems. Possible values range between 0 and 9. Higher values mean more severe problems.
Home Situations Questionnaire | Change from baseline at 1,5, 4, and 7 months
  Parents assess whether children exhibit problem behaviors in different home situations and the severity of the problems. Possible values range between 0 and 9. Higher values mean more severe problems.This measurement concerns the children who take part in the first phase of the intervention.
Attention and Executive Function Rating Inventory -Preschool | Change from baseline at 1,5, 4, and 7 months
  Early childhood education workers assess the extent to which children have problems on different areas of executive functioning (e.g. distractibility, directing and sustaining attention, planning). Possible values range between 0 and 3. Higher values mean more severe problems.

SECONDARY OUTCOMES:
Go/No-go iPad task | Change from baseline at 2 months
  A game-like task measuring response inhibition from the Early Years Toolbox. In the task, children are supposed to catch the fish and avoid the sharks. This measurement concerns children selected for the second phase of the intervention due to exhibiting difficulties in self-regulation.
Working memory iPad task | Change from baseline at 2 months
  A game-like task ("Mr. Ant") from the Early Years Toolbox. In the task, children are supposed to remember the locations of stickers placed on an ant character. This measurement concerns children selected for the second phase of the intervention due to exhibiting difficulties in self-regulation.

OTHER OUTCOMES:
Abbreviated Acceptability Rating Profile | The questionnaire is filled at 1,5 months
  Intervention providers and parents assess the acceptability of the intervention after the first phase of the intervention. Possible values range between 1 and 6. Higher values mean greater acceptability.
Abbreviated Acceptability Rating Profile | The questionnaire is filled at 4 months
  Intervention providers and parents assess the acceptability of the intervention after the second phase of the intervention. Possible values range between 1 and 6. Higher values mean greater acceptability.

CONTACTS AND LOCATIONS:
Locations (1):
- Niilo Mäki Institute, Jyväskylä, Finland